CLINICAL TRIAL: NCT06886113
Title: Effects of CorVad Percutaneous Mechanical Circulatory Support in Patients with ST Segment Elevation Myocardial Infarction Complicated by Cardiogenic Shock.
Brief Title: CorVad Myocardial Infarction Complicated with Cardiogenic Shock Trial
Acronym: Corvad AMICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_Corvad_AMICS
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cardiogenic Shock
Keywords: Acute Myocardial Infarction
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional circulatory support (Placebo Comparator): Patients randomized to conventional circulatory support
  Interventions: Device: Conventional circulatory support
- CorVad (Active Comparator): Patients randomized to CorVad
  Interventions: Device: CorVad

INTERVENTIONS:
Device: Conventional circulatory support — Control group treated with conventional circulatory support and observed in intensive care unit for a minimum of 48 hrs
  Arms: Conventional circulatory support
Device: CorVad — Control group treated with Impella CP for a minimum of 48 hrs
  Arms: CorVad

SUMMARY:
Cardiogenic shock a serious complication of a heart attack (myocardial infarction). Despite evaluation of several new treatments during the last decade, the mortality in patients with cardiogenic shock still exceeds 50%. An alternative to current management is restoration of the volume of blood pumped by the heart (cardiac output) using a ventricular assist device. In the acute setting this is difficult but can be done using the CorVad device which is a catheter-based, axial flow pump that pumps blood directly from the left ventricle into the circulation thereby restoring blood flow to the failing organs. The hypothesis of the current study is to reduce mortality and morbidity of patients with cardiogenic shock using the CorVad device. The study will be carried out as a randomized multicenter study where eligible patients will be randomized to receive conventional circulatory support or support with the CorVad device and inotropic support if needed. A total of 269 patients are planned

DETAILED DESCRIPTION:
The study is a prospective, multicenter trial in patients with AMICS randomized 1:1 to CorVad or current guideline-driven therapy with planned enrollment of 269 patients. Patients comatose after out of hospital cardiac arrest are excluded. Eligible patients are randomized immediately following shock diagnosis. Among patients randomized to receive CorVad, the device is placed prior to angioplasty. The primary endpoint is all-cause mortality at 180 days.The target population of subjects are patients with acute myocardial infarction with cardiogenic shock who need high-risk PCI treatment, and sign an informed consent form (ICF) approved by the Ethics Committee (EC). Subjects who meet the enrolment criteria as judged by the investigator will apply the trial product according to the requirements and will be followed up to 180 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. ST segment elevation myocardial infarction of less than 36 hours' duration, confirmed by new onset ST-segment elevation, or emergency angiography demonstrating acute occlusion of coronary artery, and
2. Cardiogenic shock of less than 24 hours' duration, confirmed by:

   peripheral signs of tissue hypoperfusion (arterial blood lactate ≥2.5mmol/l and/or SvO2 <55% with a normal PaO2) and systolic blood pressure less than 100mmHg and/or need for vasopressor therapy (dopamine/ norepinephrine or epinephrine), and
3. Left ventricular ejection fraction of less than 45% visually estimated or by wall motion score index >1,6.

Exclusion Criteria:

1. Shock duration N24 hours
2. Other causes of shock; hypovolemia, sepsis, pulmonary embolism or anaphylaxis
3. Shock due to mechanical complication to myocardial infarction; papillary muscle rupture, rupture of the ventricular septum or rupture of ventricular free wall.
4. Severe aorta valve regurgitation/stenosis
5. Severe peripheral arterial obstructive disease that would preclude Impella device placement
6. Mechanical aortic valve prosthesis
7. Already established mechanical circulatory support (Impella or VA-ECMO)
8. Left ventricular thrombus
9. Infective endocarditis
10. Shock due to right ventricular failure
11. Out of hospital cardiac arrest with persistent Glasgow coma scale b8 after return of spontaneous circulation. Cardiac arrest occurring in ambulance or after arrival to hospital is not an exclusion criterion.
12. Subject with documented heparin induced thrombocytopenia.
13. Life expectancy of less than 1 year due to comorbidities.
14. Mental disorder or language barrier that preclude informed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Death | up to 6 months
  Death from all causes

SECONDARY OUTCOMES:
MACCE | minimum follow-up 6 months
  Major cardiovascular and cerebrovascular events, death, cardiac transplant, escalation to permanent left ventricular assist device, re-hospitalization for heart failure
Composite saftey | up to 6 months
  Rate of major bleeding, vascular complications, and significant hemolysis
Days alive out of hospital | up to 6 months
  Days alive and out of hospital, calculated by subtracting the number of days spent in hospital, from time of randomization to end of follow-up (180 days) for each patient

OTHER OUTCOMES:
Hemodynamics | up to 7 days
  Cardiac power index
Hemodynamics | up to 7 days
  Lactate clearence
Hemodynamics | up to 7 days
  Pulmonary artery pulsatility index
Renal function | up to 30 days
  Number of Participants with acute kidney injury or need for dialysis
Bleeding | up to 30 days
  Rate of bleeding complications during admission
Revascularization strategy | During procedure
  Syntax score ( a grading system that evaluates the complexity and prognosis of patients undergoing percutaneous coronary intervention, higher scores denotes more complex disase and higher risk)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China